CLINICAL TRIAL: NCT03009825
Title: TrOma: A Cross-sectional Study Investigating Trauma Exposure, Emotion Regulation and Eating Pathology in Obese Patients
Brief Title: Trauma Exposure, Emotion Regulation and Eating Pathology in Obese Patients
Acronym: TrOma
Status: Completed | Type: Observational
Sponsor: University of Paris 5 - Rene Descartes (Other)
Collaborators: European Georges Pompidou Hospital (Other)
Responsible Party: Principal Investigator, Ruffault Alexis, Doctoral candidate, University of Paris 5 - Rene Descartes
Other Study IDs: EA4057-troma
Record Dates: First submitted 2017-01-02; First posted 2017-01-04 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Obesity
Keywords: Trauma exposure; Psychological distress; Emotion regulation; Mindfulness; Eating pathology
MeSH Terms: conditions — Obesity; Emotional Regulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the associations between lifetime exposure to traumatic events, emotion regulation strategies, and eating pathology of patients with obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Obese (BMI >= 30)
* Recruited from the nutrition service of Hôpital Européen Georges-Pompidou
* Informed consent provided

Exclusion Criteria:

* PTSD symptoms (score > 33 ; PTSD Checklist-5)
* Bariatric surgery patients
* Difficulties to understand French language
* Patients under social protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with obesity
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Self-reported binge eating pathology (BES) | Baseline
  Binge Eating Scale

SECONDARY OUTCOMES:
Self-reported anxiety and depression (HADS) | Baseline
  Hospital Anxiety and Depression Scale (2 subscales): anxiety and depression
Self-reported mindfulness skills (FFMQ) | Baseline
  Five Facets Mindfulness Questionnaire (version: 15 items): observe, describe, act with awareness, non-judgment, non-react
Self-reported emotion regulation (CERQ) | Baseline
  Cognitive Emotional Regulation Questionnaire (2 subscales): adaptive regulation and non-adaptive regulation
Self-reported eating patterns (TFEQ-R18) | Baseline
  Three Factor Eating Questionnaire (3 subscales): emotional eating, uncontrolled eating, restraint eating
Self-reported impact of traumatic event (IES-R) | Baseline
  Impact of Event Scale revised version (3 subscales): avoidance, intrusion, hyperarousal
Self-reported childhood trauma (CTQ) | Baseline
  Childhood Trauma Questionnaire (5 subscales): emotional neglect, emotional abuse, physical neglect, physical abuse, sexual abuse
Self-reported lifetime traumatic events (LEC-5) | Baseline
  Life Event Checklist (DSM-5)
Body Mass Index (kg/m2) | Baseline
  BMI as measured by a physician

OTHER OUTCOMES:
Sociodemographics and medical data | Baseline
  Form filled out by the participants

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Flahault, PhD, Study Director — University Paris 5 - Rene Descartes; Sébastien Czernichow, Pr, Principal Investigator — University Paris 5 - Rene Descartes
Locations (1):
- Hopital Europeen Georges Pompidou, Paris, France